CLINICAL TRIAL: NCT00002214
Title: Phase I Trial of S-1153 in Patients With HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexigen Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 286A; 9616T0311; 51,197
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — capravirine

INTERVENTIONS:
Drug: Capravirine

SUMMARY:
To assess the toxicity profile and determine the maximum tolerated dose (MTD), if possible, of S-1153 administered orally 3 times daily for 14 days. To investigate the clinical pharmacokinetic parameters for S-1153. To assess anti-HIV activity associated with S-1153 administration through evaluation of CD4 and viral load measurements.

DETAILED DESCRIPTION:
Two separate schedules of S-1153 are administered on this study: single dose (2 dose levels/cohorts) and repeated dose administration over 14 days (escalation through 4 dose levels/cohorts). All doses are determined by body weight.

Single-dose study (Cohort 1):

(4 patients) low-dose po, following a standardized morning meal. (4 patients) low-dose po, fasting.

Single-dose study (Cohort 2), administered during the first 3 levels of the repeated dose study and prior to the initiation of the 4th repeated dose level:

(4 patients): intermediate-dose po, following a standardized morning meal. (4 patients): intermediate-dose po, fasted. Following treatment with S-1153, all single-dose patients (Cohorts 1and 2) are observed for 21 days.

Repeated dose (escalation) study:

All doses are administered for 14 days. Three patients are entered at the starting dose of S-1153. In the absence of dose-limiting toxicity (DLT), subsequent 3-patient cohorts are entered at 3 escalating doses.

The last patient at any given dose level must be observed for 21 days prior to entry of patient at the next dose. If 1 of the initial 3 patients experiences DLT at a given level, 3 additional patients will be added at that dose; if no additional toxicity occurs, escalation resumes. If 2 or more patients at a given dose exhibit DLT, the previous dose is declared the maximum tolerated dose (MTD) and 3 additional patients (6 total) are treated at that dose.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

1. Required for patients with CD4 cell count lower than 200:

* PCP prophylaxis with aerosolized pentamidine, trimethoprim/sulfamethoxazole, mepron, or dapsone.
* Allowed:
* Continuation on an approved antiretroviral agent other than non-nucleoside reverse transcriptase inhibitors (e.g., Nevirapine) or other specifically excluded prior medications, if received without complications for at least 4 weeks prior to study entry.

Patients must have:

* Serologically documented HIV infection.
* Single-dose patients:
* CD4 cell count greater than 50 (no upper limit for single-dose cohorts). Repeated-dose patients:
* CD4 count from 50 to 500 within 35 days prior to entrance on study.
* No active opportunistic infection.

Prior Medication:

Allowed for entry onto multiple-dose study:

* Single-dose portion of S-1153 study, provided all study visits and evaluations are completed, all eligibility criteria are met, and a minimum of 30 days has elapsed before Day 1 of the repeated-dose administration.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Active opportunistic infection.

Concurrent Medication:

Excluded:

Concomitant use (within 5 half-lives prior to administration and for at least 24 hours following cessation of treatment with S-1153) of highly plasma-bound drugs with narrow therapeutic indices, including but not limited to coumadin and dilantin.

Prior Medication:

1. Investigational new drugs.

* Excluded within 30 days prior to study entry:
* Chronic (greater than 7 days) use of drugs known to affect or be extensively metabolized by cytochromes P450, including but not limited to ketoconazole, fluconazole, itraconazole, isoniazid, rifampin, rifabutin, astemizole, terfenadine, or protease inhibitors.

Prior Treatment:

Excluded within 3 weeks prior to study entry:

* Cytotoxic chemotherapy.
* Interferon treatment.
* Radiation therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Med Ctr, Boston, Massachusetts, United States